CLINICAL TRIAL: NCT04599816
Title: Levosimendan Administration in High Risk Cardiac Surgery Patients With Pulmonary Hypertension
Brief Title: Levosimendan Administration in Pulmonary Hypertension
Acronym: Levosim-PH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: annie-panagiotis
Record Dates: First submitted 2020-10-18; First posted 2020-10-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Hypertension, Pulmonary; Cardiac Failure; Pulmonary Vascular Resistance Abnormality
Keywords: pulmonary vascular resistance; pulmonary hypertension; vasodilators; cardiopulmonary bypass
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- levosimendan administration at a dose of 3 mcg/kg after anesthesia induction (Active Comparator): levosimendan will be administered at a dose of 3 mcg/kg after anesthesia induction
  Interventions: Drug: levosimendan at a dose of 3 mcg/kg
- levosimendan administration at a dose of 6 mcg/kg after anesthesia induction (Active Comparator): levosimendan will be administered at a dose of 6 mcg/kg after anesthesia induction
  Interventions: Drug: levosimendan at a dose of 6 mcg/kg
- levosimendan administration at a dose of 12 mcg/kg after anesthesia induction (Active Comparator): levosimendan will be administered at a dose of 12 mcg/kg after anesthesia induction
  Interventions: Drug: levosimendan at a dose of 12 mcg/kg

INTERVENTIONS:
Drug: levosimendan at a dose of 3 mcg/kg — levosimendan will be administered intravenously at a dose of 3 mcg/kg after anesthesia induction
  Arms: levosimendan administration at a dose of 3 mcg/kg after anesthesia induction
Drug: levosimendan at a dose of 6 mcg/kg — levosimendan will be administered intravenously at a dose of 6 mcg/kg after anesthesia induction
  Arms: levosimendan administration at a dose of 6 mcg/kg after anesthesia induction
Drug: levosimendan at a dose of 12 mcg/kg — levosimendan will be administered intravenously at a dose of 12 mcg/kg after anesthesia induction
  Arms: levosimendan administration at a dose of 12 mcg/kg after anesthesia induction

SUMMARY:
The aim of the study is to examine the pharmacokinetics and pharmacodynamic properties of Levosimendan in cardiac surgery patients with pulmonary hypertension and impaired right ventricular function.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a pathophysiological disorder hemodynamically characterized by increased pulmonary vascular resistance and pressure. This can lead to right ventricle pressure overload and failure which is worsened by cardiopulmonary bypass (CPB) and extracorporeal circulation and is accompanied by high rates of morbidity and mortality in cardiac surgery patients. Pharmacological agents used to decrease pulmonary vascular resistance and right ventricle afterload are prostaglandins, iloprost, milrinone, nitric oxide (NO) and recently Levosimendan. These agents can be administered intravenously or via inhalation.

In this study, Levosimendan will be administered in patients with pulmonary hypertension undergoing cardiac surgery. The aim of the study is to examine the pharmacokinetics and pharmacodynamic properties of Levosimendan in cardiac surgery patients with pulmonary hypertension and impaired right ventricular function. The drug will be administered in different doses to define the dose at which Levosimendan administration reduces pulmonary vascular resistance and pressure without causing significant reduction of systemic vascular resistance and pressure. The anti-inflammatory effect of the perioperative use of Levosimendan in cardiac surgery will also be studied.

In this setting, 45 patients with PH caused by left sided heart disease, will be assigned into three groups:

GROUP A: Administration of Levosimendan at a dosage of 3mcg/kg after anesthesia induction.

GROUP B: Administration of Levosimendan at a dosage of 6mcg/kg after anesthesia induction.

GROUP C: Administration of Levosimendan at a dosage of 12mcg/kg after anesthesia induction.

Before and after the administration of the drug, heart function will be evaluated by hemodynamic measurements obtained by the Swan-Ganz catheter. These parameters will be heart rate (HR), blood pressure (BP), mean pulmonary arterial pressure (MPAP), central venous pressure (CVP), cardiac output (CO), pulmonary capillary wedge pressure (PCWP), cardiac index (CI), systemic vascular resistance (SVR), pulmonary vascular resistance (PVR). Transthoracic echocardiography (TTE) and transoesophageal echocardiography (TOE) will also be used. The anti-inflammatory action of Levosimendan will also be evaluated by interleukin-6 (IL-6) measurements.

This study will lead to conclusions regarding the effectiveness of Levosimendan administration in the treatment of right heart failure and PH in cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with pulmonary hypertension due to left ventricular dysfunction based on echocardiographic diagnosis preoperatively
* elective cardiac surgery

Exclusion Criteria:

* primary pulmonary hypertension
* thromboembolic disease
* chronic obstructive pulmonary disease
* emergency surgery
* redo surgery
* inability to consent to the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
change from baseline in mean pulmonary arterial pressure (MPAP) | 20 minutes after levosimendan administration, at the end of surgery and 2 hours after Intensive Care Unit (ICU) admission
  a Swan-Ganz catheter will be used for hemodynamic measurements

SECONDARY OUTCOMES:
change from baseline in pulmonary vascular resistance (PVR) | 20 minutes after levosimendan administration, at the end of surgery and 2 hours after Intensive Care Unit (ICU) admission
  a Swan-Ganz catheter will be used for hemodynamic measurements
change from baseline in mean arterial pressure (MAP) | 20 minutes after levosimendan administration, at the end of surgery and 2 hours after Intensive Care Unit (ICU) admission
  a Swan-Ganz catheter will be used for hemodynamic measurements
change from baseline in systemic vascular resistance (SVR) | 20 minutes after levosimendan administration, at the end of surgery and 2 hours after Intensive Care Unit (ICU) admission
  a Swan-Ganz catheter will be used for hemodynamic measurements
change from baseline in pulmonary capillary wedge pressure (PCWP) | 20 minutes after levosimendan administration, at the end of surgery and 2 hours after Intensive Care Unit (ICU) admission
  a Swan-Ganz catheter will be used for hemodynamic measurements
change from baseline in cardiac output (CO) | 20 minutes after levosimendan administration, at the end of surgery and 2 hours after Intensive Care Unit (ICU) admission
  a Swan-Ganz catheter will be used for hemodynamic measurements
change from baseline in tricuspid annular plane systolic excursion (TAPSE) | 20 minutes after levosimendan administration, at the end of surgery, 2 hours after Intensive Care Unit (ICU) admission and 80 hours after levosimendan administration
  transthoracic and transesophageal echocardiography will be used for echocardiographic measurements
change from baseline in fractional area change | 20 minutes after levosimendan administration, at the end of surgery, 2 hours after Intensive Care Unit (ICU) admission and 80 hours after levosimendan administration
  transthoracic and transesophageal echocardiography will be used for echocardiographic measurements

OTHER OUTCOMES:
change from baseline in blood levels of levosimendan | 20 minutes, 6 hours, 12 hours, 24 hours and 80 hours after administration
  blood levels will be measured with liquid chromatography
change from baseline in blood levels of interleukin-6 (IL-6) | end of surgery, 6 hours, 12 hours and 24 hours after Intensive Care Unit (ICU) admission
  blood levels will be measured with the enzyme linked immunosorbent assay (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DESA, Principal Investigator — Aretaieion University Hospital
Locations (1):
- Onassis Cardiac Surgery Center, Athens, Greece

REFERENCES:
- [Background] Theodoraki K, Rellia P, Thanopoulos A, Tsourelis L, Zarkalis D, Sfyrakis P, Antoniou T. Inhaled iloprost controls pulmonary hypertension after cardiopulmonary bypass. Can J Anaesth. 2002 Nov;49(9):963-7. doi: 10.1007/BF03016884. PMID 12419726
- [Background] Theodoraki K, Thanopoulos A, Rellia P, Leontiadis E, Zarkalis D, Perreas K, Antoniou T. A retrospective comparison of inhaled milrinone and iloprost in post-bypass pulmonary hypertension. Heart Vessels. 2017 Dec;32(12):1488-1497. doi: 10.1007/s00380-017-1023-2. Epub 2017 Jul 17. PMID 28717881
- [Background] Haddad F, Couture P, Tousignant C, Denault AY. The right ventricle in cardiac surgery, a perioperative perspective: II. Pathophysiology, clinical importance, and management. Anesth Analg. 2009 Feb;108(2):422-33. doi: 10.1213/ane.0b013e31818d8b92. PMID 19151265
- [Background] Hansen MS, Andersen A, Nielsen-Kudsk JE. Levosimendan in pulmonary hypertension and right heart failure. Pulm Circ. 2018 Jul-Sep;8(3):2045894018790905. doi: 10.1177/2045894018790905. Epub 2018 Jul 6. PMID 29979110
- [Background] Boost KA, Hoegl S, Dolfen A, Czerwonka H, Scheiermann P, Zwissler B, Hofstetter C. Inhaled levosimendan reduces mortality and release of proinflammatory mediators in a rat model of experimental ventilator-induced lung injury. Crit Care Med. 2008 Jun;36(6):1873-9. doi: 10.1097/CCM.0b013e3181743e63. PMID 18496375
- [Background] Kundra TS, Nagaraja PS, Bharathi KS, Kaur P, Manjunatha N. Inhaled levosimendan versus intravenous levosimendan in patients with pulmonary hypertension undergoing mitral valve replacement. Ann Card Anaesth. 2018 Jul-Sep;21(3):328-332. doi: 10.4103/aca.ACA_19_18. PMID 30052230
- [Background] Elhassan A, Essandoh M. Inhaled Levosimendan for Pulmonary Hypertension Treatment During Cardiac Surgery: A Novel Application to Avoid Systemic Hypotension. J Cardiothorac Vasc Anesth. 2019 Apr;33(4):1169-1170. doi: 10.1053/j.jvca.2018.11.039. Epub 2018 Nov 28. No abstract available. PMID 30612930
- [Background] Zhang J, Gage EM, Ji QC, El-Shourbagy TA. A strategy for high-throughput analysis of levosimendan and its metabolites in human plasma samples using sequential negative and positive ionization liquid chromatography/tandem mass spectrometric detection. Rapid Commun Mass Spectrom. 2007;21(14):2169-76. doi: 10.1002/rcm.3046. PMID 17631672